CLINICAL TRIAL: NCT00813306
Title: A Double-blind, Randomized, Placebo-controlled, Single-centre Phase I Pharmacodynamic Cross-over Study to Assess the Effect of a Single Dose of AZD2066 Oral Solution in Comparison to Placebo on Transient Lower Esophageal Sphincter Relaxations (TLESRs) in Healthy Subjects
Brief Title: 14473 - D9126C00001 Proof of Principle Study - Effect of AZD2066 on Transient Lower Esophageal Sphincter Relaxations
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark Berner-Hansen, MD, PhDMedical Science Director, Early GI, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D9126C00001
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Reflux Episodes
Keywords: GERD; TLESR; reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — AZD2066

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- A (Experimental): AZD2066
  Interventions: Drug: AZD2066
- B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- C (Experimental): AZD2066
  Interventions: Drug: AZD2066
- D (Experimental): AZD2066
  Interventions: Drug: AZD2066
- E (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2066 — 13 mg oral solution, 1 single dose
  Arms: A
Drug: Placebo — Oral solution, 1 single dose
  Arms: B
Drug: AZD2066 — Dose to be decided after Part A, including dose A (active) and B (placebo). Oral solution, 1 single dose
  Arms: C
Drug: AZD2066 — Dose to be decided after Part A, including dose A (active) and B (placebo). Oral solution, 1 single dose
  Arms: D
Drug: Placebo — Oral solution, 1 single dose
  Arms: E

SUMMARY:
The purpose of the study is to assess the safety and tolerability of AZD2066 and to explore the effect of a single dose of AZD2066 on the function of the cardia (the opening between the stomach and the esophagus) compared to placebo (not containing any medical substance) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written consent prior to any study specific procedures.
* Healthy subjects, age 18-45 years inclusive. Females must be of no childbearing potential or must use a highly effective contraceptive method.
* Clinically normal physical findings and laboratory values at the time of pre-entry visit, as judged by the investigator.

Exclusion Criteria:

* Clinically significant illness within the 2 weeks prior to the first dose of the investigational product, including a suspected/manifested infection according to WHO risk categories 2, 3 or 4, as judged by the investigator.
* A measured LES pressure of < 5mm Hg.
* History of previous or ongoing psychiatric disease/condition.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-12; Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Manometry | 3.45 hours each study period

SECONDARY OUTCOMES:
pH | 3.45 hours each study period
Impedance | 3.45 hours each study period
Pharmacokinetic variables | 3.45 hours each study period

CONTACTS AND LOCATIONS:
Overall Officials: Marie Sundin, Study Director — AstraZeneca R&D, Mölndal, Sweden; Guy E Boeckxstaens, MD, PhD, Principal Investigator — Motiliteitscentrum (C2-310)Department of Gastroenterology,Academic Medical Centre
Locations (1):
- Research site, Amsterdam, Netherlands